CLINICAL TRIAL: NCT06995638
Title: Web-based Technology and Cognitive Training: Improving Executive Control in Cognitively Healthy Older Adults: the MUltitasking STrategy (MUST) Study
Brief Title: Improving Executive Control in Cognitively Healthy Older Adults: the MUltitasking STrategy (MUST) Study
Acronym: MUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sharon Sanz Simon, Ph.D., Assistant Professor (Principal Investigator), Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2025000330; 4R00AG078561-03 (NIH)
Record Dates: First submitted 2025-05-14; First posted 2025-05-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Aging; Alzheimer's Disease (AD)
Keywords: Aging; Cognition; Executive Functions; Randomized Controlled Trial; Cognitive Training; Neuropsychology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware of the difference between the two active conditions. Assessor will not be aware in which group condition the participant was allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strategy Training (Experimental): Participants will undergo a web-based training protocol that involves playing an online game simulating a breakfast environment, where they will perform everyday activities such as "cooking" and "setting tables" in a multitasking fashion. Participants will learn to play the game using specific strategies to optimize their performance.
  Interventions: Behavioral: Web-based Cognitive Training (with strategy)
- Regular Training (Active Comparator): Participants will undergo a web-based training protocol that involves playing an online game simulating a breakfast environment, where they will perform everyday activities such as "cooking" and "setting tables" in a multitasking fashion. Participants will learn to play the game under regular game instructions.
  Interventions: Behavioral: Web-based Cognitive Training (without strategy)
- Passive Control (No Intervention)

INTERVENTIONS:
Behavioral: Web-based Cognitive Training (with strategy) — Participants will learn to play a complex online game using specific guidance or strategy.
  Arms: Strategy Training
Behavioral: Web-based Cognitive Training (without strategy) — Participants will learn to play a complex online game without specific guidance or strategy.
  Arms: Regular Training

SUMMARY:
Developing efficient cognitive intervention for cognitively health older adults is a major public health goal, due to its potential for reducing age-related cognitive decline and Alzheimer's disease/dementia risk. Executive Control is a relevant cognitive target since it declines with aging and is critical for multi-tasking in daily life. The proposed research investigates whether playing a web-based cognitive complex game (the Breakfast Game) impacts cognitive performance in cognitively healthy older adults. To be enrolled in the study, participants will be asked to undergo a cognitive sassessment, health questionnires, and a blood exam. The intervention consist in one educational session on healthy aging, and 10 one-hour cognitive training sessions 2-3 times a week over one month. Participants will be asked to repeat the cognitive assessment within 1-2 weeks after the intervention, and after three months.

DETAILED DESCRIPTION:
The proposed research investigates whether exposure to a web-based training protocol designed to enhance executive control / multi-tasking abilities will improve cognitive performance in cognitively healthy older adults. Cognitively normal adults aged 60-75 will be randomized into three groups: 1) Web-based game with training strategy (Experimental); 2) Web-based game without training strategy (Active Control); 3) No intervention group (Passive control). Participants in groups 1 and 2 will be instructed to play the complex, high-demand online game, the Breakfast Game, for 10 one-hour sessions over 4 weeks. At study entry all participants will be asked to complete a cognitive assessment, health questionnaires, a blood exam and and education session on healthy aging. After the intervention, participants will be asked to repeat the cogntive assessment within 1-2 weeks, and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-75
* Adequate English proficiency
* Willingness to adhere to training protocol:

  * Attend 2 in-person assessments
  * Attend a blood test
  * Attend online intervention sessions and online follow-up assessment

Exclusion Criteria:

* Low test scores (below 26 on the Montreal Cognitive Assessment)
* Known history of cognitive impairment, dementia, stroke, seizure disorder, or other neuropsychiatric condition judged to impact cognitive performance.
* Taking medications known to influence cognitive performance.
* Sensory (e.g. visual, auditory) or physical (e.g. severe arthritic, orthopedic, neurologic) impairment incompatible with use of a standard computer workstation.
* Enrolled in a concurrent study that could affect the outcome of this study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the Breakfast Game scores | Training session 1, week 1; training 10, approximately 4 weeks.
  Change in the total game performance based on specific scores (number of tables and cooking scores). Higher scores represent better game outcomes.
Transfer to complex executive/attention control measure (Proximal outcome). | At baseline (week 1); post-intervention (weeks 10th to 12th); and at 3-month follow-up (week 24th)
  Alphanumeric Task score.

SECONDARY OUTCOMES:
Transfer to executive functions composite measure (Proximal outcome) | At baseline (week 1); post-intervention (weeks 10th to 12th); and at 3-month follow-up (week 24th)
  Average z-score computed with tests involving working memory, divided attention, and inhibitory control (Letter-Number, UFOV and Stroop)
Transfer to Everyday Cognition Scale (ECOG) (Distal outcome) | At baseline (week 1); post-intervention (weeks 10th to 12th); and at 3-month follow-up (week 24th)
  Scores on a scale that measures cognitive difficulties in everyday life. A higher score indicates higher levels of cognitive difficulties or change.
Transfer to Mindful Attention Awareness Scale (MAAS) (Distal outcome) | At baseline (week 1); post-intervention (weeks 10th to 12th); and at 3-month follow-up (week 24th)
  Scores on a scale that measures attention awareness. A higher score indicates higher levels of attention awareness.
Transfer to Self Efficacy for Cognitive Everyday Tasks (Distal outcome) | At baseline (week 1); post-intervention (weeks 10th to 12th); and at 3-month follow-up (week 24th)
  Scores on a scale that measures self-efficacy. A higher score indicates higher levels of self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Sanz Simon Assistant Professor, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers New Jersey Medical School, Behavior Health Sciences Building, F-Level, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in lifestyle intervention in aging.. Data or samples shared will be coded, with no private health information (PHI) included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted starting 6 months after article publication, and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the PI lab email: engaging.lab@rutgers.edu.
URL: https://sites.rutgers.edu/engaginglab/

REFERENCES:
- [Background] Blumen HM, Gopher D, Steinerman JR, Stern Y. Training cognitive control in older adults with the space fortress game: the role of training instructions and basic motor ability. Front Aging Neurosci. 2010 Nov 11;2:145. doi: 10.3389/fnagi.2010.00145. eCollection 2010. PMID 21120135
- [Background] Stern Y, Blumen HM, Rich LW, Richards A, Herzberg G, Gopher D. Space Fortress game training and executive control in older adults: a pilot intervention. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2011 Nov;18(6):653-77. doi: 10.1080/13825585.2011.613450. Epub 2011 Oct 12. PMID 21988726
- [Background] Sanz Simon S, Ben-Eliezer D, Pondikos M, Stern Y, Gopher D. Feasibility and acceptability of a new web-based cognitive training platform for cognitively healthy older adults: the breakfast task. Pilot Feasibility Stud. 2023 Aug 4;9(1):136. doi: 10.1186/s40814-023-01359-2. PMID 37542331
- See also: EngAGING Lab Website — https://sites.rutgers.edu/engaginglab/